CLINICAL TRIAL: NCT00482274
Title: Phase II Study of the Early Use of Docetaxel in Patients With Biochemical Relapse After Primary Therapy for Prostate Cancer and an Incomplete Response to Androgen Deprivation Therapy.
Brief Title: Docetaxel in Treating Patients With Relapsed Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug supplier stopped funding due to loss of study drug (docetaxel) patent.
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Tom Beer, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000546975; P30CA069533 (NIH); OHSU-2838 (Other: OHSU IRB); OHSU-SOL-06076-LM (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Results first posted 2010-08-24 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage I prostate cancer; stage II prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel

INTERVENTIONS:
Drug: docetaxel — Docetaxel 75 mg/m2 intravenously (IV) over 60 minutes will be given on day 1 of each 21 day cycle.
  Other Names: Taxotere

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well docetaxel works in treating patients with relapsed prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the complete response rate in patients with biochemically-relapsed, hormone-sensitive prostate cancer treated with docetaxel.

Secondary

* Determine the time to PSA recurrence in patients receiving this treatment.
* Determine the time to metastatic disease in patients receiving this treatment.
* Determine the time to androgen independent state in patients receiving this treatment.
* Determine the time to death from any cause in patients receiving this treatment.

OUTLINE: This is an open label study.

Patients receive docetaxel IV over 60 minutes on day 1. Treatment repeats every 21 days for 4-6 courses in the absence of unacceptable toxicity or disease progression.

After completion of study therapy, patients are followed periodically for up to 5 years.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study.

ELIGIBILITY:
Criteria for Patient eligibility

Inclusion criteria

1. Histologically confirmed adenocarcinoma of the prostate.
2. Prior primary therapy for prostate cancer, including radical prostatectomy, external beam radiation therapy, or brachytherapy.
3. Serum PSA > 0.2 ng/dL following 8 months of androgen deprivation therapy or a nadir PSA >0.2 ng/dL and at least 1 subsequent PSA values at the same or higher level, if prior to 8 months.
4. Serum testosterone < 50 ng/ml.
5. No evidence of metastases on bone scan.
6. No evidence of metastases on CT scan of the abdomen and pelvis.
7. ECOG performance status < 2.
8. Laboratory criteria for entry: absolute neutrophil count ≥ 1.2 K/cu mm, platelets ≥ 100 K/cu mm, serum bilirubin ≤ upper limit of normal (ULN), SGOT and SGPT ≤ 1.5 times institutional ULN if alkaline phosphatase ≤ ULN, alkaline phosphatase ≤ 5 times ULN if SGOT and SGPT are ≤ ULN, a serum creatinine ≤ 2 times institutional ULN.
9. Signed informed consent.

Exclusion Criteria

1. A second active malignancy during the last 5 years, except adequately treated non-melanoma skin cancer.
2. Life expectancy < 3 months.
3. Grade 2 or higher peripheral neuropathy.
4. Prior investigational agent within the past 28 days.
5. Less than a 10% decrease (or continued rise) in PSA in response to initial androgen-deprivation therapy.
6. More than 12 months since initiation of androgen-deprivation therapy.
7. Prior docetaxel chemotherapy.
8. Patients recently (within 28 days) started on corticosteroids, with the exception of inhaled and topical steroids. Patients on stable doses of systemic corticosteroids will be eligible.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz M. Beer, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - OHSU Knight Cancer Institute, Portland, Oregon
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three subjects were enrolled between 11/08 and 4/09 from the oncology clinic at OHSU. Enrollment was terminated on 11/30/09, when the sponsor withdrew funding for this study.
Groups:
- Docetaxel: Subjects received 4-6 cycles of docetaxel at 75mg/m2 every 21 days.
Period: Overall Study
Arm/Group | Docetaxel
Started | 3
Completed | 2
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Docetaxel
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (2.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Complete Response as Measured by Serum PSA Less Than 0.2 ng/ml
Description: Complete response rate, as measured by PSA and defined as a PSA ≤0.2 ng/ml in PSA-relapsed, hormone-sensitive patients treated with docetaxel.
Time Frame: While receiving study treatment (approximately 6 months)
Population: Analysis includes all subjects who completed study regimen of 6 cycles.
Measure: Number; unit: participants
Arm/Group | Docetaxel
Number analyzed (Participants) | 2
participants | 1

2. Secondary Outcome: Average Time for Participants to Develop PSA Recurrence (PSA > 0.2ng/ml)
Description: Average time for participants to develop PSA recurrence (PSA > 0.2ng/ml). Due to the limited enrollment, this analysis was not completed.
Time Frame: Average days to develop recurrence from treatment start date amount applicable participants
Population: Due to the limited enrollment, this analysis was not completed.
Arm/Group | Docetaxel
Number analyzed (Participants) | 0

3. Secondary Outcome: Time to Metastatic Disease
Description: Due to the limited enrollment, this analysis was not completed.
Time Frame: Measured at Time of documented metastases (no historical estimate is available)
Population: Due to limited enrollment, this analysis was not completed
Arm/Group | Docetaxel
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Androgen Independent State
Description: Due to the limited enrollment, this analysis was not completed.
Time Frame: Measured at date of documented androgen independence (no estimate available)
Population: Due to the limited enrollment, this analysis was not completed.
Arm/Group | Docetaxel
Number analyzed (Participants) | 0

5. Secondary Outcome: Time to Death From Any Cause
Description: Due to the limited enrollment, this analysis was not completed.
Time Frame: measured at date of death (no estimate available)
Population: Due to the limited enrollment, this analysis was not completed.
Arm/Group | Docetaxel
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Docetaxel
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel (N=3)
Fatigue (General disorders) | 2 (2)
alopecia (General disorders) | 1 (1)
pain (General disorders) | 1 (1)
insomnia (General disorders) | 1 (1)
hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
watering eyes (Eye disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to withdrawal of sponsor support, this study was terminated after only 3 subjects were enrolled (of the planned 36 subjects). Sufficient data were not obtained to make statistically significant conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No